CLINICAL TRIAL: NCT04532905
Title: Energy Expenditure During Acute and Chronic Resistance Exercises in Healthy Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University (Other)
Collaborators: Taipei Medical University Hospital (Other)
Responsible Party: Principal Investigator, Chih-Wei, Peng, Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: N202004023
Record Dates: First submitted 2020-07-10; First posted 2020-08-31 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Healthy
Keywords: Strength training; Normal population; energy expenditure

STUDY DESIGN:
Intervention Model Description: The study will include two groups: 1) control (untrained) and 2) strength training (trained)
Who Masked: Participant
Masking Description: Only participants will be masked for group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- without previous strength training experience (Sham Comparator): control (untrained) group will receive intervention as five exercises: dumbbell bent row over, dumbbell deadlift, dumbbell lunge. dumbbell shoulder press, and dumbbell squat
  Interventions: Other: Strength Training Exercises Therapy
- with previous strength training experience (Experimental): experimental (trained) group will receive intervention as five exercises: dumbbell bent row over, dumbbell deadlift, dumbbell lunge. dumbbell shoulder press, and dumbbell squat
  Interventions: Other: Strength Training Exercises Therapy

INTERVENTIONS:
Other: Strength Training Exercises Therapy — Five type of exercises: dumbbell bent row over, deadlift, lunge, shoulder press, and squat with each three sets and 10 repetitions. Between each set there will be 2-3 minute rest period and 8-10 minute rest period among each exercise type.

SUMMARY:
The present study aims to predict energy expenditure models for some resistance training exercises like: dumbbell bent row over, dumbbell deadlift, dumbbell lunge, dumbbell shoulder press, and dumbbell squat using oxygen consumption or Metabolic Equivalents (METs) as a dependent variable while blood pressure, heart rate, respiratory exchange ratio, blood lactate, rate of perceived exertion, body mass index, body weight, body height, body fat composition, muscle strength, and surface electromyography of selected muscles as independent variables. The previous literature measures energy expenditure for various lower and upper body resistance training exercises but it devoid for dumbbell bent row over, dumbbell deadlift, dumbbell lunge, dumbbell shoulder press, and dumbbell squat energy expenditure models between untrained and trained participants. The subject will come for 5-8 times clinical trial for total 10-20 days. After the completion of this study, the participant will know about their energy expenditure during included strength training exercises.

DETAILED DESCRIPTION:
The present study aims to predict energy expenditure models for some resistance training exercises like: dumbbell bent row over, dumbbell deadlift, dumbbell lunge, dumbbell shoulder press, and dumbbell squat using oxygen consumption or Metabolic Equivalents (METs) as a dependent variable while blood pressure, heart rate, respiratory exchange ratio, blood lactate, rate of perceived exertion, body mass index, body weight, body height, body fat composition, muscle strength, and surface electromyography of selected muscles as independent variables. The previous literature measures energy expenditure for various lower and upper body resistance training exercises but it devoid for dumbbell bent row over, dumbbell deadlift, dumbbell lunge, dumbbell shoulder press, and dumbbell squat energy expenditure models between untrained and trained participants. The subject will come for 5-8 times clinical trial for total 10-20 days. After the completion of this study, the participant will know about their energy expenditure during included strength training exercises.

The study will include total 30 participants; 15 normal healthy young individuals and 15 athletes with regular resistance exercise training experience. The experiments will be divided into 2 stages. The first stage experiment will be conducted in 10 young individuals into two groups. The group one (untrained) will include 5 normal healthy individuals without resistance exercise training experience and group two (trained) will include 5 individuals with regular resistance training experience of two months. The second stage will proceed more 20 young participants (10 participants in each group) to determine the resistance exercise energy expenditure.

ELIGIBILITY:
Inclusion Criteria:

* Male and female young healthy participants and athletes having strength training experience minimum of 2 months
* Skeletally mature, between 20-40 years of age.
* Able to understand and comply with study requirements
* Able to understand and give informed consent.
* Not having any metabolic, systematic, musculoskeletal disease or injury
* No recent surgical procedure which can hinder exercise training
* Not taking medication especially sedatives, anti-depressant, or anti-hypertensive etc
* Physically fit according to Physical Activity Readiness Questionnaire (Par-Q)

Exclusion Criteria:

* Age below 20 or above 40
* Having any metabolic, systematic, musculoskeletal disease or injury
* Recent surgical procedure

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — To conduct a study on male and female participants
Enrollment: 30 (Estimated)
Dates: Start 2020-07-06 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
oxygen consumption (VO2) | VO2 data will be processed for resting stage of 2-10 minutes before the start of exercise.
  VO2 will be recorded through cortex metalyzer breath by breath during exercises. There will be data recording for rest period of 2-10 minutes before the start of exercise.
oxygen consumption (VO2) | VO2 data will be processed for each set of exercise 1. Day 1 to up to 3-4 weeks (for exercise 1)
  VO2 will be recorded through cortex metalyzer breath by breath during exercises. The data will be recorded during each exercise 1 (Dumbbell Bent Row Over). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks.
oxygen consumption (VO2) | VO2 data will be processed for each set of exercise 2. Day 1 to up to 3-4 weeks (for exercise 2)
  VO2 will be recorded through cortex metalyzer breath by breath during exercises. The data will be recorded during each exercise 2 (Dumbbell Deadlift). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks.
oxygen consumption (VO2) | VO2 data will be processed for each set of exercise 3. Day 1 to up to 3-4 weeks (for exercise 3)
  VO2 will be recorded through cortex metalyzer breath by breath during exercises. The data will be recorded during each exercise 3 (Dumbbell Lunge). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks.
oxygen consumption (VO2) | VO2 data will be processed for each set of exercise 4. Day 1 to up to 3-4 weeks (for exercise 4)
  VO2 will be recorded through cortex metalyzer breath by breath during exercises. The data will be recorded during each exercise 4 (Dumbbell Shoulder Press). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks.
oxygen consumption (VO2) | VO2 data will be processed for each set of exercise 5. Day 1 to up to 3-4 weeks (for exercise 5)
  VO2 will be recorded through cortex metalyzer breath by breath during exercises. The data will be recorded during each exercise 5 (Dumbbell Squat). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks.
Heart rate | Heart rate data will be processed for resting stage of 2-10 minutes before the start of exercise.
  Heart rate will be recorded through ECG electrodes during exercises. There will be data recording for rest period of 2-10 minutes before the start of exercise.
Heart rate | Heart rate data will be processed for each set of exercise 1. Day 1 to up to 3-4 weeks (for exercise 1)
  Heart rate will be recorded through ECG electrodes during exercises. The data will be recorded during each exercise 1 (Dumbbell Bent Row Over). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks.
Heart rate | Heart rate data will be processed for each set of exercise 2. Day 1 to up to 3-4 weeks (for exercise 2)
  Heart rate will be recorded through ECG electrodes during exercises. The data will be recorded during each exercise 2 (Dumbbell Deadlift). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks.
Heart rate | Heart rate data will be processed for each set of exercise 3. Day 1 to up to 3-4 weeks (for exercise 3)
  Heart rate will be recorded through ECG electrodes during exercises. The data will be recorded during each exercise 3 (Dumbbell Lunge). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks.
Heart rate | Heart rate data will be processed for each set of exercise 4. Day 1 to up to 3-4 weeks (for exercise 4)
  Heart rate will be recorded through ECG electrodes during exercises. The data will be recorded during each exercise 4 (Dumbbell Shoulder Press). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks.
Heart rate | Heart rate data will be processed for each set of exercise 5. Day 1 to up to 3-4 weeks (for exercise 5)
  Heart rate will be recorded through ECG electrodes during exercises. The data will be recorded during each exercise 5 (Dumbbell Squat). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks.
Respiratory Exchange Ratio (RER) | RER data will be processed for resting stage of 2-10 minutes before the start of exercise.
  RER will be recorded through cortex metalyzer. There will be data recording for rest period of 2-10 minutes before the start of exercise.
Respiratory Exchange Ratio (RER) | RER data will be processed for each set of exercise 1. Day 1 to up to 3-4 weeks (for exercise 1)
  RER will be recorded through cortex metalyzer breath by breath during exercises. The data will be recorded during each exercise 1 (Dumbbell Bent Row Over). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks
Respiratory Exchange Ratio (RER) | RER data will be processed for each set of exercise 2. Day 1 to up to 3-4 weeks (for exercise 2)
  RER will be recorded through cortex metalyzer breath by breath during exercises. The data will be recorded during each exercise 2 (Dumbbell Deadlift). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks
Respiratory Exchange Ratio (RER) | RER data will be processed for each set of exercise 3. Day 1 to up to 3-4 weeks (for exercise 3)
  RER will be recorded through cortex metalyzer breath by breath during exercises. The data will be recorded during each exercise 3 (Dumbbell Lunge). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks
Respiratory Exchange Ratio (RER) | RER data will be processed for each set of exercise 4. Day 1 to up to 3-4 weeks (for exercise 4)
  RER will be recorded through cortex metalyzer breath by breath during exercises. The data will be recorded during each exercise 4 (Dumbbell Shoulder Press). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks
Respiratory Exchange Ratio (RER) | RER data will be processed for each set of exercise 5. Day 1 to up to 3-4 weeks (for exercise 5)
  RER will be recorded through cortex metalyzer breath by breath during exercises. The data will be recorded during each exercise 5 (Dumbbell Squat). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks
surface electromyography | Surface electromyography data will be processed for each set of exercise 1. Day 1 to up to 3-4 weeks (for exercise 1)
  It will be measured by Noraxon surface electromyography (sEMG) sensors over pectoralis major, latissimus dorsi, hamstrings, quadriceps, erector spinae, or deltoid of both sides. The data will be recorded during each exercise 1 (Dumbbell Bent Row Over). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks.
surface electromyography | Surface electromyography data will be processed for each set of exercise 2. Day 1 to up to 3-4 weeks (for exercise 2)
  It will be measured by Noraxon surface electromyography (sEMG) sensors over pectoralis major, latissimus dorsi, hamstrings, quadriceps, erector spinae, or deltoid of both sides. The data will be recorded during each exercise 2 (Dumbbell Deadlift). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks.
surface electromyography | Surface electromyography data will be processed for each set of exercise 3. Day 1 to up to 3-4 weeks (for exercise 3)
  It will be measured by Noraxon surface electromyography (sEMG) sensors over pectoralis major, latissimus dorsi, hamstrings, quadriceps, erector spinae, or deltoid of both sides. The data will be recorded during each exercise 3 (Dumbbell Lunge). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks.
surface electromyography | Surface electromyography data will be processed for each set of exercise 4. Day 1 to up to 3-4 weeks (for exercise 4)
  It will be measured by Noraxon surface electromyography (sEMG) sensors over pectoralis major, latissimus dorsi, hamstrings, quadriceps, erector spinae, or deltoid of both sides. The data will be recorded during each exercise 4 (Dumbbell Shoulder Press). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks.
surface electromyography | Surface electromyography data will be processed for each set of exercise 5. Day 1 to up to 3-4 weeks (for exercise 5)
  It will be measured by Noraxon surface electromyography (sEMG) sensors over pectoralis major, latissimus dorsi, hamstrings, quadriceps, erector spinae, or deltoid of both sides. The data will be recorded during each exercise 5 (Dumbbell Squat). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks.
Blood pressure | Blood pressure data during resting stage of exercise will be used before the start of exercise.
  Sphygmomanometer will be used (systolic and diastolic) to record blood pressure. There will be data recording during rest before the start of exercise.
Blood pressure | Blood pressure data value for exercise 1 will be used. Day 1 to up to 3-4 weeks (for exercise 1)
  Sphygmomanometer will be used (systolic and diastolic) to record blood pressure. The data will be recorded within 5 minutes of exercise 1 (Dumbbell Bent Row Over). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks.
Blood pressure | Blood pressure data value for exercise 2 will be used. Day 1 to up to 3-4 weeks (for exercise 2)
  Sphygmomanometer will be used (systolic and diastolic) to record blood pressure. The data will be recorded within 5 minutes of exercise 2 (Dumbbell Deadlift). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks.
Blood pressure | Blood pressure data value for exercise 3 will be used. Day 1 to up to 3-4 weeks (for exercise 3)
  Sphygmomanometer will be used (systolic and diastolic) to record blood pressure. The data will be recorded within 5 minutes of exercise 3 (Dumbbell Lunge). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks.
Blood pressure | Blood pressure data value for exercise 4 will be used. Day 1 to up to 3-4 weeks (for exercise 4)
  Sphygmomanometer will be used (systolic and diastolic) to record blood pressure. The data will be recorded within 5 minutes of exercise 4 (Dumbbell Shoulder Press). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks.
Blood pressure | Blood pressure data value for exercise 5 will be used. Day 1 to up to 3-4 weeks (for exercise 5)
  Sphygmomanometer will be used (systolic and diastolic) to record blood pressure. The data will be recorded within 5 minutes of exercise 5 (Dumbbell Squat). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks.
Blood lactate level | Blood lactate data during resting stage of exercise will be used before the start of exercise.
  Blood lactate will be recorded through lactate meter. There will be data recording during rest before the start of exercise.
Blood lactate level | Blood lactate data value for exercise 1 will be used. Day 1 to up to 3-4 weeks (for exercise 1)
  Blood lactate will be recorded through lactate meter. The data will be recorded after 5 minutes of exercise 1 (Dumbbell Bent Row Over). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks.
Blood lactate level | Blood lactate data value for exercise 2 will be used. Day 1 to up to 3-4 weeks (for exercise 2)
  Blood lactate will be recorded through lactate meter. The data will be recorded after 5 minutes of exercise 2 (Dumbbell Deadlift). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks.
Blood lactate level | Blood lactate data value for exercise 3 will be used. Day 1 to up to 3-4 weeks (for exercise 3)
  Blood lactate will be recorded through lactate meter. The data will be recorded after 5 minutes of exercise 3 (Dumbbell Lunge). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks.
Blood lactate level | Blood lactate data value for exercise 4 will be used. Day 1 to up to 3-4 weeks (for exercise 4)
  Blood lactate will be recorded through lactate meter. The data will be recorded after 5 minutes of exercise 4 (Dumbbell Shoulder Press). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks.
Blood lactate level | Blood lactate data value for exercise 5 will be used. Day 1 to up to 3-4 weeks (for exercise 5)
  Blood lactate will be recorded through lactate meter. The data will be recorded after 5 minutes of exercise 5 (Dumbbell Squat). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks.
Rate of perceived exertion (RPE) | RPE score during resting stage of exercise will be used before the start of exercise.
  The RPE score will be recorded before the start of training session.
Rate of perceived exertion (RPE) | RPE score for exercise 1 will be used. Day 1 to up to 3-4 weeks (for exercise 1)
  The RPE will be recorded within 5 minutes of exercise 1 (Dumbbell Bent Row Over). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks.
Rate of perceived exertion (RPE) | RPE score for exercise 2 will be used. Day 1 to up to 3-4 weeks (for exercise 2)
  The RPE will be recorded within 5 minutes of exercise 2 (Dumbbell Deadlift). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks.
Rate of perceived exertion (RPE) | RPE score for exercise 3 will be used. Day 1 to up to 3-4 weeks (for exercise 3)
  The RPE will be recorded within 5 minutes of exercise 3 (Dumbbell Lunge). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks.
Rate of perceived exertion (RPE) | RPE score for exercise 4 will be used. Day 1 to up to 3-4 weeks (for exercise 4)
  The RPE will be recorded within 5 minutes of exercise 4 (Dumbbell Shoulder Press). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks.
Rate of perceived exertion (RPE) | RPE score for exercise 5 will be used. Day 1 to up to 3-4 weeks (for exercise 5)
  The RPE will be recorded within 5 minutes of exercise 5 (Dumbbell Squat). Each exercise will consist of three sets of 30-40 seconds. And each set will be of 10 repetition (3-4 second per repetition). Each subject will receive 3-6 training sessions for up to 3-4 weeks.

SECONDARY OUTCOMES:
Physical fitness status | baseline before start of exercise
  Physical activity readiness questionnaire will be used. This questionnaire assesses baseline fitness level of participants. It has two options either ''yes'' or ''no'' in explaining the basic seven fitness related questions. The more the questions have ''yes'' answers meaning participant health status is not good and they are not eligible for this study. The other category of questions evaluate existence of any medical condition with ''yes'' or ''no'' options which can exclude participant from this study.
Body mass index (BMI) | baseline before start of exercise and after all three or six training sessions for up to 3-4 weeks.
  body composition measuring scale will be used. The body composition will be measured two times during the study before the start of training and after three or six training sessions for up to 3-4 weeks. The weight will be measured in kilogram (kg) and height in meters (m) to report BMI in kg/m^2. The change in body composition will be compared before and after all training sessions.
Body fat percentage | baseline before start of exercise and after all three or six training sessions for up to 3-4 weeks.
  Body fat will be measured with measuring scale. The body fat will be measured two times during the study before the start of training and after three or six training sessions for up to 3-4 weeks. The change in body fat percentage will be compared before and after all training sessions.
Muscle Strength | baseline before start of exercise and after all three or six training sessions for up to 3-4 weeks.
  Hand held dynamometer will be used for the same muscles pectoralis major, latissimus dorsi, hamstrings, quadriceps, erector spinae, or deltoid of both sides. The strength will be measured two times during the study before the start of training and after three or six training sessions for up to 3-4 weeks. The change in muscle strength will be compared before and after all training sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baechle, T. R., & Earle, R. W. (2008). Essentials of strength training and conditioning: Human kinetics.
- [Background] Thompson, W. R., Gordon, N. F., & Pescatello, L. S. (2010). ACSM's guidelines for exercise testing and prescription: Lippincott Williams & Wilkins.
- [Background] Lambert MI, Borresen J. Measuring training load in sports. Int J Sports Physiol Perform. 2010 Sep;5(3):406-11. doi: 10.1123/ijspp.5.3.406. PMID 20861529
- [Background] Scott CB, Croteau A, Ravlo T. Energy expenditure before, during, and after the bench press. J Strength Cond Res. 2009 Mar;23(2):611-8. doi: 10.1519/JSC.0b013e31818c2845. PMID 19197214
- [Background] Benito PJ, Alvarez-Sanchez M, Diaz V, Morencos E, Peinado AB, Cupeiro R, Maffulli N; PRONAF Study Group. Cardiovascular Fitness and Energy Expenditure Response during a Combined Aerobic and Circuit Weight Training Protocol. PLoS One. 2016 Nov 10;11(11):e0164349. doi: 10.1371/journal.pone.0164349. eCollection 2016. PMID 27832062
- [Background] Phillips WT, Ziuraitis JR. Energy cost of the ACSM single-set resistance training protocol. J Strength Cond Res. 2003 May;17(2):350-5. doi: 10.1519/1533-4287(2003)0172.0.co;2. PMID 12741877

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-22): https://cdn.clinicaltrials.gov/large-docs/05/NCT04532905/Prot_SAP_001.pdf